CLINICAL TRIAL: NCT01696318
Title: Management Models for Cardiovascular Risk Reduction in Primary for Brazil: Developing a Program for Cardiovascular Prevention and Randomized Clinical Trial
Brief Title: Program for Cardiovascular Prevention and Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Federal University of Rio Grande do Sul (Other)
Collaborators: Hospital Moinhos de Vento (Other)
Responsible Party: Principal Investigator, Fabiana Viegas Raimundo, PhD, Federal University of Rio Grande do Sul
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: U1111-1134-6977; HMV - 680 (Other: Comite de Ética em Pesquisa Hospital Moinhos de Vento)
Record Dates: First submitted 2012-09-22; First posted 2012-10-01 (Estimated); Last update posted 2016-01-15 (Estimated); Status verified 2016-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Palliative Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Educational program (No Intervention): Educational Program with Professional Physical Education, Pharmacist and Nutritionist
- Educational program and individual care (Experimental): Educational program and individual care with professional Physical Education; Pharmacist and Nutritionist
  Interventions: Behavioral: Support for the Family Health Team

INTERVENTIONS:
Behavioral: Support for the Family Health Team — Participation in physical educator, dietitian and pharmacist in primary health care
  Arms: Educational program and individual care

SUMMARY:
Develop and evaluate a model of organization and management in the management of patients with cardiovascular risk factors (hypertension, diabetes mellitus, smoking, obesity, physical inactivity, dyslipidemia and family history) in primary care aimed at the compliance, control and treatment effectiveness.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of hypertension (> 140/90 mmHg)
* Age > 40 years
* Sitting: USF da Restinga e Extremo Sul - USF Chapéu do Sol and USF Paulo Viaro

Exclusion Criteria:

* Institutionalized individuals
* Patients with mental illness or disabling chronic illnesses
* Users of health services belonging to the supplementary health
* Individuals with life expectancy less than 1 year

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 256 (Actual)
Dates: Start 2012-05; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Blood Pressure | Change from baseline in Systolic Blood Pressure at 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Carisi Polanczyc, PhD, Study Director — UFRGS/HMV
Locations (1):
- Hospital Moinhos de Vento, Porto Alegre, Rio Grande do Sul, Brazil

REFERENCES:
- [Derived] Kuhmmer R, Lazzaretti RK, Guterres CM, Raimundo FV, Leite LE, Delabary TS, Caon S, Bastos GA, Polanczyk CA. Effectiveness of multidisciplinary intervention on blood pressure control in primary health care: a randomized clinical trial. BMC Health Serv Res. 2016 Aug 31;16(1):456. doi: 10.1186/s12913-016-1703-0. PMID 27581760